CLINICAL TRIAL: NCT00926094
Title: Prevalence of Impaired Glucose Tolerance (IGT) in Patients With Frozen Shoulder
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Ori Safran, Hadassah Medical Organization
Other Study IDs: SAF04-HMO-CTIL
Record Dates: First submitted 2009-06-21; First posted 2009-06-23 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-04

CONDITIONS: Frozen Shoulder; Impairment Glucose Tolerance
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- 1
- 2

SUMMARY:
Idiopathic Adhesive Capsulitis, Frozen Shoulder is a condition in which there is a limitation and significant pain at the shoulder and it is increases with shoulder movements. The causes are not clear. The prevalence of this condition is four times higher in diabetic patient compare to the general population.

The relation between frozen shoulder and impaired glucose tolerance remain unclear.

Our hypothesis is that patients with no diabetes and that suffer from frozen shoulder have a higher prevalence of impaired glucose tolerance than the general population age matched.

ELIGIBILITY:
Inclusion Criteria:

1. age 30-60.
2. previous Xray that eliminates other disease of the shoulder.
3. previous US that eliminates tendon shoulder rupture
4. shoulder movement in all directions, with limitation in the external rotation (at least 50%)

Exclusion Criteria:

1. Diagnosed Diabetes (pregnancy diabetes includes)
2. Taking Hyperglycemic medications (like Steroids)
3. Fracture or operation in the shoulder before the diagnosis of frozen shoulder.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: people that were diagnosed with frozen shoulder at the last three years and are not diabetic.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel